CLINICAL TRIAL: NCT02606955
Title: Probing the Dry Weight (DW) by Bioimpedance (BIA): Which is the Gold Standard Between Clinical DW and BIA DW?
Brief Title: Probing the Dry Weight by Bioimpedance: The Resistance Stabilization Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miulli General Hospital (Other)
Responsible Party: Principal Investigator, Carlo Basile, M.D., Scientific Director of the Division of Nephrology, Miulli General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REST./COLLABORATIVE STUDY
Record Dates: First submitted 2015-10-08; First posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Uremia
Keywords: Bioimpedance; Dry weight; Hemodialysis; Resistance
MeSH Terms: conditions — Uremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIA REST (Experimental): BIA DW assessment
  Interventions: Device: BIA DW

INTERVENTIONS:
Device: BIA DW — All patients undergo a Clinical DW assessment. Then, they undergo a HD session in which BIA DW (injection of 800 microAmpere at 50 kilohertz alternating sinusoidal current with a standard tetrapolar technique) is determined. BIA DW is determined by performing the REsistance Stabilization Test (REST).
  Other Names: BIA Resistance Stabilization Test (REST)

SUMMARY:
Clinical methods are fundamental in probing the DW. They must be supported by strict BIA protocols. REST appears to be a (the) brilliant solution in solving the old problem of DW in HD patients

DETAILED DESCRIPTION:
Probing the dry weight (DW) was largely dependent on clinical subjective estimates until recently. New bedside non-invasive tools have been developed with the aim of providing more objective information on volume status and guiding physicians in the quest for DW. Among them, bioimpedance (BIA) appears to be very promising.

Very recently, a BIA test aimed at assessing DW in hemodialysis (HD) patients has been developed, the "REsistance Stabilization Test" (REST). It is called BIA DW. Its rationale is based on the achievement of the flattening of the curve of the ratio R0/Rt (R0 is resistance at time 0 and Rt is resistance at a given time t during the HD session) of less than + 1% over 20 minutes in the presence of ongoing ultrafiltration.

Study protocol: the Clinical DW is the gold standard by definition. It is determined under strict clinical surveillance by the same attending physician. She/he will be helped by a clinical score of volume state about symptoms and signs of hypo- or hypervolemia. Then, this Clinical DW will be compared with BIA DW, as obtained after performing REST

ELIGIBILITY:
Inclusion Criteria

* stable uremic patients
* thrice weekly hemodialysis treatment
* start of hemodialysis treatment since at least 3 months

Exclusion Criteria

* overt edema
* liver cirrhosis
* cardiac failure
* serum albumin < 3g/dl
* pregnancy
* metallic implants or a pacemaker
* limb amputation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the gold standard method for the measurement of DW (in kg) through the comparison of clinical DW (as determined by means of a validated clinical score) and BIA DW (measurement of the resistance in kilohertz). | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Basile, MD, Principal Investigator — Mulli General Hospital
Locations (2):
- Italy (2):
  - Nephrology and dialysis unit Miulli General Hospital, Acquaviva delle Fonti, Bari
  - Divisionof Nephrology, Solofra

REFERENCES:
- [Background] Basile C, Libutti P, Lisi P, Rossi L, Lomonte C. Probing the dry weight by bioimpedance: the resistance stabilization test. J Nephrol. 2015 Aug;28(4):517-20. doi: 10.1007/s40620-014-0159-8. Epub 2014 Dec 6. PMID 25480486